CLINICAL TRIAL: NCT04780438
Title: Dapagliflozin to Prevent Atrial Fibrillation Recurrence After Transcatheter Pulmonary Venous Isolation.
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: G.Gennimatas General Hospital (Other)
Collaborators: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Ioannis Anagnostopoulos, MD, G.Gennimatas General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2662
Record Dates: First submitted 2021-03-02; First posted 2021-03-03 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Atrial Fibrillation Recurrent; Pulmonary Venous Isolation; Catheter Ablation; Sodium-glucose Co-transporter 2 Inhibitors
Keywords: dapagliflozin; Sodium-glucose co-transporter 2 inhibitors; Atrial Fibrillation; recurrence; catheter ablation; SGLT2 inhibitors
MeSH Terms: conditions — Atrial Fibrillation; Recurrence | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin (Active Comparator): Patients who will be randomized to receive dapagliflozin following catheter ablation.
  Interventions: Drug: Dapagliflozin
- Placebo (Placebo Comparator): Patients who will be randomized to receive placebo following catheter ablation.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Patients rendomized in this arm will receive dapagliflozin at a target dose of 10mg once daily.
  Arms: Dapagliflozin
Drug: Placebo — Patients rendomized in this arm will receive placebo.
  Arms: Placebo

SUMMARY:
Transcatheter left atrial antral ablation, aiming at complete electrical isolation of the pulmonary veins (PVI), has become mainstay in atrial fibrillation (AF) treatment. This approach has been proved superior to medical rhytmh control strategy in maintaining sinus rhythm. Moreover PVI has been associated with significant survival benefit in patients with heart failure and reduced left ventricular ejection fraction. Nevertheless, despite progress in the field of catheter ablation, recurrence rates remain high.

Inhibitors of type 2 sodium- glucose co-transporter (SGLT2i) is a relatively recent addition to the array of anti-diabetic agents, becoming part of everyday clinical practice. However, although SGLT2i were first used solely as antidiabetics because of their glycosuric effect, further research demonstrated that these drugs may independently reduce cardiovascular events, especially in patients with heart failure, a benefit that was consistent among diabetic and non-diabetic patients. Moreover, pleiotropic effects have been observed, including a reno-protective action.

These findings suggest that SGLT2i mechanisms of action extend beyond the obvious increase in urinary sodium and glucose excretion. Various studies propose that these drugs promote favourable metabolic changes in myocardial energetics, while they also inhibit inflamation and sympathetic activation, resulting in restriction of induced fibrosis and structural remodeling, which are key elements in atrial fibrillation generation and maintenance.

These findings suggest that the use of SGLT2i could offer antiarrhythmic benefit by reducing and/or reversing structural and electrical remodeling, leading to the assumption that use of theese drugs could reduce recurrences after transcatheter AF ablation.

ELIGIBILITY:
Inclusion Criteria:

Age>18 years Atrial Fibrillation (paroxysmal or sustained); Written informed consent; Glomerular Filtration Rate (GFR) >45 ml/min/1.73m2 (Cockroft-Gault equation)

Exclusion Criteria:

Hypertrophic cardiomyopathy (Left ventricular wall thickness ≥15mm, not explained by abnormal pressure/volume conditions); Severe mitral valve stenosis (as defined in European Guidelines); Active malignancy; Participation in other intervention studies; Pregnancy or willing of pregnancy during the follow up period Guideline Class I or equivalent indication for treatment with a SGLT2 inhibitor

*Eligible patients randomized in the active comparator arm will be also included in a prospective observational registry study regarding the role of SGLT2 inhibitors in post-ablation AF recurrence.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of survival free of AF/ atrial tachycardia (AT) recurrence between the two study arms. | 18 months from the PVI procedure
  AF/AT are defined as any episodes of AF or atrial flutter or other re-entrant atrial tachycardia recorded either on surface ECG or on Holter monitoring and lasting for at least 30 s. All episodes will be reviewed by two independent electrophysiologists, who will be blinded as to patient identity and randomization.The first 3 months after the ablation procedure will be regarded as a blanking period.

OTHER OUTCOMES:
Incidence (cases per 100 patient-years) of hypoglycemia in both arms | 18 months from the PVI procedure
  Any episode of hypoglycemia defined as serum glucose 60< mg/dl associated with symptoms of hypoglycemia.
Incidence (cases per 100 patient-years)of diabetic ketoacidosis | 18 months from the PVI procedure
  Any episode of metabolic acidosis (pH<7.3) with decreased serum bicarbonate (<18mEq/ml) and increased anion gap (>10) and increased serum glucose (>250mg/dl) and positive urine dipstick test for ketones.
Incidence (cases per 100 patient-years)of lower urinary tract infections | 18 months from the PVI procedure
Comparison of all cause mortality between the two groups | 18 months from the PVI procedure

CONTACTS AND LOCATIONS:
Overall Officials: Spyridon Deftereos, MD, Principal Investigator — 2nd Department of Cardiology, National and Kapodistrian University of Athens, Faculty of Medicine, Athens, Greece
Locations (2):
- Greece (2):
  - Cardiology Department, Athens General Hospital "G. Gennimatas", Athens, Greece, Athens
  - 2nd Department of Cardiology, National and Kapodistrian University of Athens, Faculty of Medicine, Athens, Greece., Athens

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Haissaguerre M, Jais P, Shah DC, Takahashi A, Hocini M, Quiniou G, Garrigue S, Le Mouroux A, Le Metayer P, Clementy J. Spontaneous initiation of atrial fibrillation by ectopic beats originating in the pulmonary veins. N Engl J Med. 1998 Sep 3;339(10):659-66. doi: 10.1056/NEJM199809033391003. PMID 9725923
- [Result] Asad ZUA, Yousif A, Khan MS, Al-Khatib SM, Stavrakis S. Catheter Ablation Versus Medical Therapy for Atrial Fibrillation: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Circ Arrhythm Electrophysiol. 2019 Sep;12(9):e007414. doi: 10.1161/CIRCEP.119.007414. Epub 2019 Aug 21. PMID 31431051
- [Result] Packer DL, Mark DB, Robb RA, Monahan KH, Bahnson TD, Poole JE, Noseworthy PA, Rosenberg YD, Jeffries N, Mitchell LB, Flaker GC, Pokushalov E, Romanov A, Bunch TJ, Noelker G, Ardashev A, Revishvili A, Wilber DJ, Cappato R, Kuck KH, Hindricks G, Davies DW, Kowey PR, Naccarelli GV, Reiffel JA, Piccini JP, Silverstein AP, Al-Khalidi HR, Lee KL; CABANA Investigators. Effect of Catheter Ablation vs Antiarrhythmic Drug Therapy on Mortality, Stroke, Bleeding, and Cardiac Arrest Among Patients With Atrial Fibrillation: The CABANA Randomized Clinical Trial. JAMA. 2019 Apr 2;321(13):1261-1274. doi: 10.1001/jama.2019.0693. PMID 30874766
- [Result] Ganesan AN, Shipp NJ, Brooks AG, Kuklik P, Lau DH, Lim HS, Sullivan T, Roberts-Thomson KC, Sanders P. Long-term outcomes of catheter ablation of atrial fibrillation: a systematic review and meta-analysis. J Am Heart Assoc. 2013 Mar 18;2(2):e004549. doi: 10.1161/JAHA.112.004549. PMID 23537812
- [Result] Zinman B, Wanner C, Lachin JM, Fitchett D, Bluhmki E, Hantel S, Mattheus M, Devins T, Johansen OE, Woerle HJ, Broedl UC, Inzucchi SE; EMPA-REG OUTCOME Investigators. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2117-28. doi: 10.1056/NEJMoa1504720. Epub 2015 Sep 17. PMID 26378978
- [Result] Wiviott SD, Raz I, Bonaca MP, Mosenzon O, Kato ET, Cahn A, Silverman MG, Zelniker TA, Kuder JF, Murphy SA, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Ruff CT, Gause-Nilsson IAM, Fredriksson M, Johansson PA, Langkilde AM, Sabatine MS; DECLARE-TIMI 58 Investigators. Dapagliflozin and Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2019 Jan 24;380(4):347-357. doi: 10.1056/NEJMoa1812389. Epub 2018 Nov 10. PMID 30415602
- [Result] Neal B, Perkovic V, Mahaffey KW, de Zeeuw D, Fulcher G, Erondu N, Shaw W, Law G, Desai M, Matthews DR; CANVAS Program Collaborative Group. Canagliflozin and Cardiovascular and Renal Events in Type 2 Diabetes. N Engl J Med. 2017 Aug 17;377(7):644-657. doi: 10.1056/NEJMoa1611925. Epub 2017 Jun 12. PMID 28605608
- [Result] McMurray JJV, Solomon SD, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Sabatine MS, Anand IS, Belohlavek J, Bohm M, Chiang CE, Chopra VK, de Boer RA, Desai AS, Diez M, Drozdz J, Dukat A, Ge J, Howlett JG, Katova T, Kitakaze M, Ljungman CEA, Merkely B, Nicolau JC, O'Meara E, Petrie MC, Vinh PN, Schou M, Tereshchenko S, Verma S, Held C, DeMets DL, Docherty KF, Jhund PS, Bengtsson O, Sjostrand M, Langkilde AM; DAPA-HF Trial Committees and Investigators. Dapagliflozin in Patients with Heart Failure and Reduced Ejection Fraction. N Engl J Med. 2019 Nov 21;381(21):1995-2008. doi: 10.1056/NEJMoa1911303. Epub 2019 Sep 19. PMID 31535829
- [Result] Packer M, Anker SD, Butler J, Filippatos G, Pocock SJ, Carson P, Januzzi J, Verma S, Tsutsui H, Brueckmann M, Jamal W, Kimura K, Schnee J, Zeller C, Cotton D, Bocchi E, Bohm M, Choi DJ, Chopra V, Chuquiure E, Giannetti N, Janssens S, Zhang J, Gonzalez Juanatey JR, Kaul S, Brunner-La Rocca HP, Merkely B, Nicholls SJ, Perrone S, Pina I, Ponikowski P, Sattar N, Senni M, Seronde MF, Spinar J, Squire I, Taddei S, Wanner C, Zannad F; EMPEROR-Reduced Trial Investigators. Cardiovascular and Renal Outcomes with Empagliflozin in Heart Failure. N Engl J Med. 2020 Oct 8;383(15):1413-1424. doi: 10.1056/NEJMoa2022190. Epub 2020 Aug 28. PMID 32865377
- [Result] Zannad F, Ferreira JP, Pocock SJ, Anker SD, Butler J, Filippatos G, Brueckmann M, Ofstad AP, Pfarr E, Jamal W, Packer M. SGLT2 inhibitors in patients with heart failure with reduced ejection fraction: a meta-analysis of the EMPEROR-Reduced and DAPA-HF trials. Lancet. 2020 Sep 19;396(10254):819-829. doi: 10.1016/S0140-6736(20)31824-9. Epub 2020 Aug 30. PMID 32877652
- [Result] Heerspink HJL, Stefansson BV, Correa-Rotter R, Chertow GM, Greene T, Hou FF, Mann JFE, McMurray JJV, Lindberg M, Rossing P, Sjostrom CD, Toto RD, Langkilde AM, Wheeler DC; DAPA-CKD Trial Committees and Investigators. Dapagliflozin in Patients with Chronic Kidney Disease. N Engl J Med. 2020 Oct 8;383(15):1436-1446. doi: 10.1056/NEJMoa2024816. Epub 2020 Sep 24. PMID 32970396
- [Result] Lopaschuk GD, Verma S. Mechanisms of Cardiovascular Benefits of Sodium Glucose Co-Transporter 2 (SGLT2) Inhibitors: A State-of-the-Art Review. JACC Basic Transl Sci. 2020 Jun 22;5(6):632-644. doi: 10.1016/j.jacbts.2020.02.004. eCollection 2020 Jun. PMID 32613148
- [Result] Verma S, McMurray JJV. SGLT2 inhibitors and mechanisms of cardiovascular benefit: a state-of-the-art review. Diabetologia. 2018 Oct;61(10):2108-2117. doi: 10.1007/s00125-018-4670-7. Epub 2018 Aug 22. PMID 30132036
- [Result] Andreadou I, Efentakis P, Balafas E, Togliatto G, Davos CH, Varela A, Dimitriou CA, Nikolaou PE, Maratou E, Lambadiari V, Ikonomidis I, Kostomitsopoulos N, Brizzi MF, Dimitriadis G, Iliodromitis EK. Empagliflozin Limits Myocardial Infarction in Vivo and Cell Death in Vitro: Role of STAT3, Mitochondria, and Redox Aspects. Front Physiol. 2017 Dec 19;8:1077. doi: 10.3389/fphys.2017.01077. eCollection 2017. PMID 29311992
- [Result] Wan N, Rahman A, Hitomi H, Nishiyama A. The Effects of Sodium-Glucose Cotransporter 2 Inhibitors on Sympathetic Nervous Activity. Front Endocrinol (Lausanne). 2018 Jul 26;9:421. doi: 10.3389/fendo.2018.00421. eCollection 2018. PMID 30093883
- [Result] Maejima Y. SGLT2 Inhibitors Play a Salutary Role in Heart Failure via Modulation of the Mitochondrial Function. Front Cardiovasc Med. 2020 Jan 8;6:186. doi: 10.3389/fcvm.2019.00186. eCollection 2019. PMID 31970162
- [Result] Li WJ, Chen XQ, Xu LL, Li YQ, Luo BH. SGLT2 inhibitors and atrial fibrillation in type 2 diabetes: a systematic review with meta-analysis of 16 randomized controlled trials. Cardiovasc Diabetol. 2020 Aug 26;19(1):130. doi: 10.1186/s12933-020-01105-5. PMID 32847602